CLINICAL TRIAL: NCT02614651
Title: Prospective Pilot Study on the Quantitative Evaluation of Vision Parameters Needed by Virtual Reality Goggle Displays for Subjects With Concentric Visual Field Constriction. AUgmented REality for the Visually Impaired - Part 1
Brief Title: AUgmented REality for the Visually Impaired - Part 1
Acronym: AUREVI 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LOCAL/2015/IMGD-01; 2016-A00099-42 (Other: RCB number)
Record Dates: First submitted 2015-11-19; First posted 2015-11-25 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2016-05

CONDITIONS: Retinitis Pigmentosa; Glaucoma
MeSH Terms: conditions — Retinitis Pigmentosa; Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The study population (Experimental): The study population consists of subjects with a concentric constriction of the visual field (retinitis pigmentosa, glaucoma) whose motor capacity allows the use of a computer keyboard with one hand. Subjects are recruited on a voluntary basis, from information disseminated to professionals in the rehabilitation of functional low vision and patient associations, in the Ophthalmology Service of the University Hospital of Nimes and within the ARAMAV Institute.
  Intervention: Find visual comfort threshold related to light intensity
  Intervention: Find the size of the visual field
  Intervention: Effectiveness of brightness control
  Intervention: Performance of color correction
  Intervention: Vuzix Wrap 1200DX virtural reality glasses
  Interventions: Procedure: Find visual comfort threshold related to light intensity; Procedure: Find the size of the visual field; Procedure: Effectiveness of brightness control; Procedure: Performance of color correction; Device: Vuzix Wrap 1200DX virtural reality glasses

INTERVENTIONS:
Procedure: Find visual comfort threshold related to light intensity — In this testing session, the patient's visual comfort threshold related to light intensity will be determined. Test sessions are kept under 45 minutes.
  The subject is sitting in front of a keyboard and a computer screen. He/she is invited to recognize letters successively displayed in the center of the screen, this center is marked with a black cross. Each letter appearance is preceded by a beep. The subject must click on the "space" bar on the keyboard as soon as he/she recognizes the letter, then gives his/her answer orally.
Procedure: Find the size of the visual field — For these tests, the subject is seated at a table, 1.5m from a wall. It features a computer keyboard. It projects an image on the wall, using to a video projector. An image moving towards a target (along 16 different trajectories) is used to evaluate the size of the visual field.
Procedure: Effectiveness of brightness control — During this testing session, the investigators seek to evaluate the effectiveness of the algorithms used to control the brightness.
  The subject is in a room with four different computers. The subject is asked to identify the objects displayed on different computer monitors in the room: he/she must press a key on the keyboard when he/she detects an object and state aloud the nature of the object.
Procedure: Performance of color correction — During this session, the investigators try to assess the performance for the color vision correction (saturation and hue).
  The subject, while wearing the virtual reality glasses + camera performs a test (twice) that requires matching colored dots (i.e. a Farnsworth test) under controlled light conditions.
Device: Vuzix Wrap 1200DX virtural reality glasses — The other interventions are performed with the use of virtual reality glasses, specifically the Vuzix Wrap 1200DX. In case of technical difficulties, the latter can be swapped with the Oculus Rift model or another model. The associated webcameras are from Logitech, and the exact model used can vary and does not carry any importance for this research.

SUMMARY:
The main objective of this study is to quantify vision parameters in subjects with concentric visual field constriction, and this in relation to the display on virtual reality goggles. More specifically:

* The maximum brightness value for visual comfort (THRESHOLD_MAX)
* The minimum value of the perceptible light contrast in low light perceptible (THRESHOLD_MIN)
* The speed of light change adaptation in the range [THRESHOLD_MAX-THRESHOLD_MIN] and [THRESHOLD_MIN-THRESHOLD_MAX].

DETAILED DESCRIPTION:
Secondary objectives are to:

A. Quantifying the device parameters "RV glasses + camera" depending on visual acuity and the visual field of each subject:

* Optimal extent of the visual field provided by the device "RV glasses + camera".

B. Measuring the effectiveness of different image processing algorithms used in the development of the software part of this technical assist device:

* Capture and display HDR images (High Dynamic Range)
* Color adjustment.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The subject is suffering from retinitis pigmentosa or glaucoma with concentric visual field constriction and presents with:
* An acuity in the better eye superior or equal to 1/10 in near vision,
* A binocular field of between 1° and 30°,
* A good central fixation, absence of central scotoma,
* Motor capability for using a computer keyboard with one hand.

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, or under guardianship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* Subjects with (or evolving toward) a multiple sensory disability, or one including cognitive disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-05; Primary Completion 2017-04-20 (Actual); Study Completion 2017-05-29 (Actual)

PRIMARY OUTCOMES:
The maximum brightness value for visual comfort (THRESHOLD_MAX) | 0 to 6 months
The minimum value of the perceptible light contrast in low light perceptible (THRESHOLD_MIN) | 0 to 6 months
The speed of light change adaptation within a pre-specified range (getting dimmer) | 0 to 6 months
  The pre-specified range goes from THRESHOLD_MAX down to THRESHOLD_MIN.
The speed of light change adaptation within a pre-specified range (getting brighter) | 0 to 6 months
  The pre-specified range goes from THRESHOLD_MIN up to THRESHOLD_MAX.

SECONDARY OUTCOMES:
Optimal range (in degrees) of the visual field provided by the device "RV glasses + camera" | 0 to 6 months
Response time in seconds | 0 to 6 months
Number of correct responses | 0 to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Marc, PhD, Study Director — Laboratoire LGI2P, Ecole Nationale Supérieure des Mines; Luc Jeanjean, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHRU de Nîmes - Hôpital Universitaire Carémea, Nîmes, France